CLINICAL TRIAL: NCT03333681
Title: Evaluation of Mesenchymal Stem Cell Therapy Effects on the Cellular and Humoral Immune Responses and Additionally Study on the Effect of Chemokines in Homing of the Immune Cells in Refractory Rheumatoid Arthritis Patients
Brief Title: Evaluation of Stem Cell Therapy Effects on the Immune Response in Rheumatoid Arthritis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Mojgan Mohammadi, Associate professor, Mashhad University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 931523; 122 (Other Grant/Funding Number: Council for Stem Cell Sciences and Technologies)
Record Dates: First submitted 2017-09-14; First posted 2017-11-07 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Stem Cells; Cellular immunity; Humoral immunity; chemokines; homing of immune cells
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Refractory rheumatoid arthritis patients (Experimental): Autologous mesenchymal stem cells
  Interventions: Biological: Autologous mesenchymal stem cells

INTERVENTIONS:
Biological: Autologous mesenchymal stem cells — A single intravenous administration of autologous bone marrow derived mesenchymal stem cells(1000000 to 2000000 cells/Kg)

SUMMARY:
1. Objectives: Evaluation of mesenchymal stem cell therapy effects on cellular and humoral immune responses in refractory rheumatoid arthritis (RA) patients.
2. Design: This study has been performed as a phase 1 clinical trial.
3. Setting and conduct: Autologous bone marrow derived mesenchymal stem cells were obtained by bone marrow aspiration and cultured in Minimum Essential Medium-Alpha (MEM-alpha) for 4 weeks in standard clean room and then transfused to RA patients intravenously.
4. Participant's major eligibility criteria is as follows: Ten refractory rheumatoid arthritis patients who show resistance to non biological Disease-modifying antirheumatic drugs (DMARDs) after 6 to 12 months have been enrolled in this study.
5. Intervention: A single dose of intravenous autologous bone marrow derived mesenchymal stem cells have been administered into patients with resistance to non-biological DMARDs.
6. Main outcome measures (variables): Finding of mesenchymal stem cell therapy effects on the cellular and humoral immune responses and evaluation of the effect of chemokines in homing of immune cells following the intervention.

DETAILED DESCRIPTION:
Refractory rheumatoid arthritis patients who met the inclusion/exclusion criteria have been selected. After signing informed consent form, autologous stem cells were obtained by bone marrow aspiration. Isolation and culture (3 to 4 weeks in MEM-alpha medium) of mesenchymal stem cells (MSCs) were performed in accredited good manufacturing practices (GMP) clean room. A panel of cluster of differentiation (CD) markers including CD105, CD166, CD44, CD45, CD90, and CD34 were checked for making sure about differentiation of cells into MSCs after 3-4 weeks of cell culture. Viability of MSCs was checked by Trypan blue testing and all of the cultivations were negative for bacterial contamination. A single dose of 1000000 to 2000000 mesenchymal stem cells/kg infused into patients intravenously. To prevent anaphylactic reactions, a single intravenous dose of hydrocortison (100 ml) and oral dimenhydrinate (10 ml) were administered before MSCs infusion into patients. The effects of mesenchymal stem cells on the cellular and humoral immune responses and also the role of chemokines in homing of immune cells were studied at time points 1, 6 and 12 months after intravenous administration of MSCs in refractory rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Resistant RA patients to non-biological DMARDs;
* Treated RA patients by non-biological drugs;
* Treated RA patients by Prednisolone, Hydroxychloroquine, Sulfasalazine and Methotrexate;
* Patients age between 35-60 years;
* Refractory RA patients with no other rheumatologic disorders and inflammatory diseases.

Exclusion Criteria:

* Non-resistant RA patients to non-biological DMARDs.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 15 (Estimated)
Dates: Start 2016-06-20 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Effect of mesenchymal stem cells therapy on the percentage of regulatory T cells | At 0 and 6 months follow up
  Percentage change in regulatory T cells from baseline which is analysed by fluorescence-activated cell sorting (FACS)

CONTACTS AND LOCATIONS:
Overall Officials: Mojgan Mohammadi, Ph.D, Principal Investigator — Mashhad University of Medical Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alvaro-Gracia JM, Jover JA, Garcia-Vicuna R, Carreno L, Alonso A, Marsal S, Blanco F, Martinez-Taboada VM, Taylor P, Martin-Martin C, DelaRosa O, Tagarro I, Diaz-Gonzalez F. Intravenous administration of expanded allogeneic adipose-derived mesenchymal stem cells in refractory rheumatoid arthritis (Cx611): results of a multicentre, dose escalation, randomised, single-blind, placebo-controlled phase Ib/IIa clinical trial. Ann Rheum Dis. 2017 Jan;76(1):196-202. doi: 10.1136/annrheumdis-2015-208918. Epub 2016 Jun 7. PMID 27269294
- [Background] Liang J, Li X, Zhang H, Wang D, Feng X, Wang H, Hua B, Liu B, Sun L. Allogeneic mesenchymal stem cells transplantation in patients with refractory RA. Clin Rheumatol. 2012 Jan;31(1):157-61. doi: 10.1007/s10067-011-1816-0. Epub 2011 Aug 12. PMID 21837432
- [Background] Wang L, Wang L, Cong X, Liu G, Zhou J, Bai B, Li Y, Bai W, Li M, Ji H, Zhu D, Wu M, Liu Y. Human umbilical cord mesenchymal stem cell therapy for patients with active rheumatoid arthritis: safety and efficacy. Stem Cells Dev. 2013 Dec 15;22(24):3192-202. doi: 10.1089/scd.2013.0023. Epub 2013 Oct 4. PMID 23941289
- [Derived] Rahimi Khorashad M, Ghoryani M, Gowhari Shabgah A, Shariati-Sarabi Z, Tavakkol Afshari J, Mohammadi M. The Effects of Mesenchymal Stem Cells on the Gene Expression of TGF-beta and IFN-gamma in Patients with Rheumatoid Arthritis. Iran J Allergy Asthma Immunol. 2023 Apr 30;22(2):183-189. doi: 10.18502/ijaai.v22i2.12679. PMID 37496411